CLINICAL TRIAL: NCT06849219
Title: Comparison of Oxcarbazepine Versus Carbamazepine in the Management of Trigeminal Neuralgia in Patients Presenting in Outpatient Department of Neurology in Jinnah Postgraduate Medical Centre
Brief Title: Comparison of Oxcarbazepine Versus Carbamazepine in the Management of Trigeminal Neuralgia
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Rizwana Malahat Ahmad, Postgraduate Trainee, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO.F.2-81/2024-GENL/77/JPMC
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal neuralgia; Carbamazepine; Oxcarbazepine
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Oxcarbazepine; Carbamazepine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxcarbazepine (Group A) (Experimental): Starting dose of oxcarbazepine 150 mg BD, titrated up if no pain relief
  Interventions: Drug: Oxcarbazepine
- Carbamazepine (Group B) (Active Comparator): Starting dose of carbamazepine 100 mg BD, titrated up if no relief
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Oxcarbazepine — Oxcarbazepine will be started at a dose of 150 mg BD, and follow-up will be done every month. Dose will be titrated up if minimal pain relief, to a maximum dose of 1800 mg per day.
  Other Names: Telox; Trioptal; Oxalepsy
  Arms: Oxcarbazepine (Group A)
Drug: Carbamazepine — Carbamazepine will be started at a dose of 100 mg BD, and follow-up will be done every month. Dose will be titrated up if minimal pain relief, to a maximum dose of 1200 mg per day.
  Other Names: Tegral; Seizunil; Teril
  Arms: Carbamazepine (Group B)

SUMMARY:
Trigeminal neuralgia is a debilitating neurological condition, affecting quality of life in most affected patients. Carbamazepine has traditionally been used for the management of this condition, but it has a moderate effectiveness and a poor side-effect profile. Oxcarbazepine is more tolerable, and has a more favorable side-effect profile. This study aims to compare the effectiveness of oxcarbazepine and carbamazepine in the management of this condition, for improved prescription practices in the future.

DETAILED DESCRIPTION:
INTRODUCTION:

According to the International Headache Society, Trigeminal neuralgia is defined as "a disorder characterized by recurrent unilateral brief electric shock-like pain, abrupt in onset and termination, limited to the distribution of one or more divisions of the trigeminal nerve and triggered by innocuous stimuli" [1]. The trigeminal nerve (V) is the fifth and largest of all cranial nerves, and it is responsible for detecting sensory stimuli that arise from the craniofacial area including the forehead, cheek, and lower jaw [2]. It is a highly debilitating disorder that impacts on basic human functions such as talking, eating, drinking and touching the face, thereby resulting in a poor quality of life [3, 4].

Trigeminal neuralgia is considered a rare condition, affecting 4 to 13 people per 100,000 people annually. Women are more commonly affected than men. The female-to-male prevalence ratio ranges from 1.5 to 1.7 to 1. Most cases of trigeminal neuralgia occur after age 50, but the disease may be seen in the second and third decades of life; trigeminal neuralgia is rarely diagnosed in childhood. The lifetime prevalence of trigeminal neuralgia in population-based studies is estimated at 0.16% to 0.3% [5, 6]. A Pakistani study by Usman J, et al. audited the trigeminal neuralgia patients visiting the tertiary care hospital over a period of two years and reported a 0.46% prevalence of trigeminal neuralgia [7].

Trigeminal neuralgia is usually suspected through historical, physical and clinical examination findings. These patients should undergo neuroimaging with magnetic resonance imaging (MRI) and magnetic resonance angiography (MRA) whenever possible for confirmation of trigeminal neuralgia [6, 8, 9]. Medical therapy is the preferred initial therapeutic intervention for patients with trigeminal neuralgia. The antiepileptics carbamazepine or oxcarbazepine are the preferred initial therapeutic agents [10]. Carbamazepine is FDA indicated for epilepsy, trigeminal neuralgia, and acute manic and mixed episodes in bipolar I disorder [11]. Oxcarbazepine is an analogue of carbamazepine and is often used in acute orofacial pain episodes lasting seconds, as well as in the trigeminal nerve and its branches. Oxcarbazepine is preferred over carbamazepine because it has advantages over carbamazepine and lesser negative effects [12]. A study by Iqbal S, et al was conducted on efficacy of carbamazepine and oxcarbazepine for treating trigeminal neuralgia and reported a complete response in 42.9% of patients with carbamazepine and 67.9% of patients with oxcarbazepine. Frequency of adverse effects was higher for carbamazepine as that of Oxcarbazepine. i.e. 35.7% vs. 14.3% [13]. Another study by Di Stefano G, et al. reported that the initial proportion of responders was 88.3% with carbamazepine, and 90.9% with oxcarbazepine. Side effects occurred more frequently in patients treated with carbamazepine (43.6%) than with oxcarbazepine (30.3%) [14].

The rationale of the study is to compare the efficacy of oxcarbazepine and carbamazepine in the management of trigeminal neuralgia in patients presenting in the outpatient department of neurology at Jinnah Postgraduate Medical Centre. International and local data is very scarce regarding the comparisons of both of these drugs for treating trigeminal neuralgia. However, the effects of these drugs have been documented in the literature in comparison to other drugs or as a triple therapy combination. So, taking both drugs as monotherapy for treating trigeminal neuralgia can lead us to conclude which drug is superior as a monotherapy so that, in the future, drug with better efficacy will be preferred. The results of the study will be helpful in the selection of an appropriate and more effective drug for the treatment of trigeminal neuralgia.

OBJECTIVE:

To compare the efficacy of oxcarbazepine and carbamazepine in the management of trigeminal neuralgia in patients presenting in outpatient department of neurology Jinnah Postgraduate Medical Centre.

OPERATIONAL DEFINITION:

1. TRIGEMINAL NEURALGIA:

   It will be confirmed by using International Classification of Headache Disorders edition 3 (ICHD-3) diagnostic criteria.

   Diagnostic Criteria:

   Recurrent paroxysms of unilateral facial pain in the distribution(s) of one or more divisions of the trigeminal nerve, with no radiation beyond, and fulfilling criteria B and C.

   A. Pain has all of the following characteristics: lasting from a fraction of a second to 2 minutes, severe intensity and electric shock-like, shooting, stabbing or sharp in quality.

   B. Precipitated by innocuous stimuli within the affected trigeminal distribution.

   C. Not better accounted for by another ICHD-3 diagnosis.
2. VISUAL ANALOGUE SCALE (VAS)

   VAS is a tool used to measure pain, with 0 indicating no pain and 10 indicating the worst pain. Pain intensity on the VAS is divided as follows:
   * 0 for no pain.
   * 1-3 for mild pain.
   * 4-6 for moderate pain.
   * 7-10 for severe pain.
3. EFFICACY The effectiveness of both drugs will be measured by the frequency of pain attacks.

   * Good Response: No attacks of pain.
   * Average Response: Two to three attacks of pain per day.
   * Nonresponsive: No decrease in the frequency of attacks of pain.
4. SAFETY Safety of patient will be assessed on presence of side effects such as drowsiness (feeling sleepy or tired during the day time), dizziness (feeling faint, weak or unsteady), diplopia (double vision), nausea (feeling to vomit), and hyponatremia (serum sodium level < 135 mEq/L).

HYPOTHESIS:

* Null Hypothesis: There is no difference in the efficacy of Oxcarbazepine and carbamazepine in the management of trigeminal neuralgia.
* Alternative Hypothesis: Oxcarbazepine is more effective than carbamazepine in the management of trigeminal neuralgia.

MATERIAL AND METHODS:

SETTING:

This study will be conducted at Ward 28, Department of Neurology Jinnah Postgraduate Medical Centre (JPMC) Karachi.

DURATION OF STUDY:

Six months

STUDY DESIGN:

Randomized controlled trial.

SAMPLE SIZE:

The sample size calculation was done by using the "Open Epi" software for sample size calculation by using the proportion of Iqbal S, et al. who reported a complete response in 42.9% of patients with carbamazepine and 67.9% of patients with oxcarbazepine [13], by taking confidential interval 95% and power 80%. Calculated sample size was 122 (61 in each group).

* Group A (oxcarbazepine) = 61 patients
* Group B (carbamazepine) = 61 patients

SAMPLING TECHNIQUE:

Non-probability consecutive sampling technique.

DATA COLLECTION PROCEDURE:

This study will be performed after the permission of Research evaluation unit (REU) of College of Physicians and Surgeons Pakistan (CPSP) and written informed consent for the study will be obtained from the patient who fulfill the inclusion criteria.

Outpatient visiting Ward 28 of Neurology Department Jinnah Postgraduate Medical Centre, Karachi and who fulfills the inclusion criteria will be included in the study. Detailed demographic details of each patient including name, gender, age, residence, educational status and employment status will be obtained. Each patient will be assessed for duration of pain, severity of pain, frequency of pain and side of pain. After that each patient will be assessed for pain severity by using the VAS. Each patient will be asked to point out the number on VAS that best represents the intensity of their pain.

Patients will be randomly distributed to either Group A (oxcarbazepine) or Group B (carbamazepine) using a lottery method. Group A patients will be treated with oxcarbazepine (150 mg twice daily up to 1800 mg) and Group B patients will be treated with carbamazepine (100 mg twice daily up to 1200 mg). Dose will depends on severity of symptoms. Patients will be counseled about presence of side effects such as drowsiness, dizziness, diplopia, nausea and hyponatremia, and instructed to report to principal investigator in case of side effects causing any disability or interference in daily activities. Each patient will be followed up every month and the final outcome i.e., the efficacy of the treatment will be assessed six months after the treatment. All results will be collected and filled in proforma accordingly by the researcher.

DATA ANALYSIS PROCEDURE:

After collection of data the analyses will be conducted by using Statistical Package for Social Science (SPSS) software, Version 25.

Mean and standard deviation will be calculated for quantitative variables like age (years), duration of pain (days) and frequency of pain before and after treatment, VAS pain score before and after treatment in both groups. Frequency and percentages will be calculated for categorical variables like gender, age in groups, residence, educational status, employment status, side of pain, severity of pain before and after treatment, safety and efficacy of treatment in both groups. Efficacy will be compared between the group by applying chi-square test. Effect modifiers like gender, age in groups, residence, educational status, employment status, duration of pain in groups and side of pain will be controlled by stratification. Post-stratification chi-square test will be applied by taking p value ≤ 0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender (male or female)
* Patients of age 25-80 years
* Patients presenting with trigeminal neuralgia of any frequency and severity (according to operational definition) for six months
* Patients not already receiving carbamazepine or oxcarbazepine for the management of trigeminal neuralgia

Exclusion Criteria:

* Patients who have undergone any surgical procedure for the treatment of trigeminal neuralgia
* Patients with renal and hepatic issue such as chronic renal failure and chronic liver disease
* Patients not already receiving carbamazepine or oxcarbazepine for the management of trigeminal neuralgia
* Patients with seizures
* Patients who are intolerant to and allergic to both treatment drugs (oxcarbazepine and carbamazepine)
* Pregnant and Iactating mothers
* Patients who are not willing to participate in the study

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Improvement in pain scores | 6 months
  Visual analog scale (score from 0 to 10, where 10 indicates worst pain)

SECONDARY OUTCOMES:
Adverse effects of drugs in both arms | 6 months
  Common side-effects will be asked about at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rizwana Malahat Ahmad, MBBS, Principal Investigator — Jinnah Postgraduate Medical Centre
Locations (1):
- Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No